CLINICAL TRIAL: NCT01017588
Title: Lumbar Support for Low Back Pain Prevention in Rubber Tapper
Brief Title: PSU Lumbar Support for Prevention of Low Back Pain in Rubber Tapper
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Boonsin Tangtrakulwanich, Department of Orthopaedic surgery, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC52-200-11-4-2
Record Dates: First submitted 2009-11-17; First posted 2009-11-20 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Low Back Pain
Keywords: lumbar support; rubber tapper
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- back exercise (Experimental): strengthening back exercise
  Interventions: Device: PSU lumbar back support

INTERVENTIONS:
Device: PSU lumbar back support — wear PSU back supprt during doing rubber tapper

SUMMARY:
This study aims to evaluate the efficacy of lumbar support for low back pain prevention in rubber tapper. The investigators will randomized the participants(rubber tapper) into 2 groups;lumbar support and no support.The participant will be instructed for brace use. The sample size required are 200 subjects with 100 in each group. The subject will be evaluated every 3 month for the incidence of low back pain and quality of life after using the support.

ELIGIBILITY:
Inclusion Criteria:

* current rubber tapper

Exclusion Criteria:

* underlying rheumatologic condition
* previous significant low back pain
* previous back surgery

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
incidence of low back pain | 6 month, 1 and 2 years

SECONDARY OUTCOMES:
Roland Moris score | 6 month, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD.,Ph.D., Principal Investigator — Department of Orthopaedic Surgery, Faculty of Medicine, Prince of Songkla University, Hat Yai, Songkhla, Thailand
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand